CLINICAL TRIAL: NCT04080427
Title: Effects of THC on Retention of Memory for Fear Extinction Learning in PTSD: R33 Study
Brief Title: Effects of Delta9-tetrahydrocannabinol (THC) on Retention of Memory for Fear Extinction Learning in PTSD: R33 Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Christine Rabinak, PhD, Associate Professor & Principal Investigator, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: R33MH111935 (NIH); R61MH111935 (NIH)
Record Dates: First submitted 2019-08-30; First posted 2019-09-06 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Posttraumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Sugars; Dronabinol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo capsule (Placebo Comparator): In a randomized, double-blind, placebo-controlled, between-subjects design, the investigators will administer a single oral dose of dronabinol (7.5mg) or placebo (PBO) approximately two hours prior to each weekly exposure session (up to 9 sessions) in a standard prolonged exposure treatment protocol comprising 12 session overall.
  Half of the participants will receive 7.5mg dronabinol (n=50) and the other half of the participants will receive placebo (n=50).
  Interventions: Drug: Placebo capsule
- Dronabinol 7.5 milligram oral capsule (Experimental): In a randomized, double-blind, placebo-controlled, between-subjects design, the investigators will administer a single oral dose of dronabinol (7.5mg) or placebo (PBO) approximately two hours prior to each weekly exposure session (up to 9 sessions) in a standard prolonged exposure treatment protocol comprising 12 session overall.
  Half of the participants will receive 7.5mg dronabinol (n=50) and the other half of the participants will receive placebo (n=50).
  Interventions: Drug: Dronabinol 7.5 milligram oral capsule

INTERVENTIONS:
Drug: Placebo capsule — Placebo is administered just prior to weekly exposure sessions by the oral route and contains only dextrose in opaque capsules.
  Other Names: sugar pill
  Arms: Placebo capsule
Drug: Dronabinol 7.5 milligram oral capsule — Dronabinol (7.5mg) is administered just prior to weekly exposure sessions by the oral route and is placed in an opaque capsule with dextrose filler.
  Other Names: Marinol
  Arms: Dronabinol 7.5 milligram oral capsule

SUMMARY:
The goal of this study is to look at how a type of drug called cannabinoids are related to the processing of fear signals, the experience of emotions and fear, and the pattern of activity in the brain that is involved in these processes and how this relates to the treatment of post-traumatic stress disorder (PTSD). PTSD is an anxiety disorder that occurs after experiencing a traumatic event(s) and is characterized by unwanted memories of the trauma(s) through flashbacks or nightmares, avoidance of situations that remind the person of the event, difficulty experiencing emotions, loss of interest in activities the person used to enjoy, and increased arousal, such as difficulty falling asleep or staying asleep, anger and hypervigilance. The information gained from this study could lead to the development of new treatments for persons who suffer from anxiety or fear-based disorders.

DETAILED DESCRIPTION:
The total time commitment estimated per participant 18 study visits. This is broken down below:

Visit 1: Questionnaires, Screening, and Orientation: During this visit the potential participant will learn about the study procedures, sign the informed consent documents, and fill out a packet of forms that ask about his or her race and ethnic background, use of drugs and alcohol and physical and mental health.

Visit 2: Pre-Treatment Behavioral Tests and and Magnetic Resonance (MR) Scan: During this visit the participant will complete several computer tasks, and the study staff will be measuring reaction time and psychophysiological measures.The tasks that the participant will perform will show three different images and an aversive stimulus (e.g. loud burst of noise or animated snake) may follow one image most of the time, while the other images may never be followed by the aversive cue. The participant will need to try to predict whether the aversive cue will occur or not based on which image is shown and will be asked to repeatedly rate on a scale how likely it is that he or she thinks an aversive cue will occur after each image. Lastly, during the session the participant will also be asked to report his or her level of anxiety on a scale from 0 to 100.

Visit 3: Pre-Treatment Behavioral Tests and MR Scan: This visit will be very similar to Visit 2. Participants will participate in the same type of task inside the MR scanner, while the study staff measures reaction time and psychophysiological responding and brain activation. Participants will view the same images he or she did previously, and may experience the same aversive stimulus as during Visit 2. Participants will again be asked to rate how much they expect to experience the aversive stimulus after each image and will also be asked to report their level of anxiety on a scale from 0 to 100.

Visits 4 & 5: Prolonged Exposure (PE) Sessions 1 & 2: These sessions will consist of psychoeducation that includes discussion or reactions to trauma , treatment rationale, breathing retraining, and review of SUDS to assess level of distress from 0 to 100 (100=extreme anxiety/distress) when facing fears. One session occurs weekly across 2 weeks.

Visits 6-14: PE Sessions 3-11: These sessions will consist of repeated exposures to trauma memories (imaginal exposure) and avoided situations (in vivo exposure). As is standard, patients will also practice exposures (e.g., listen to tapes of imaginal exposure, carry out in vivo exposure) outside of PE sessions as "homework". At exposure-focused sessions (Sessions 3-11) either THC or PBO will be administered just before the session. One session occurs weekly across 8 weeks.

Visit 15: PE Session 12 [Post-treatment Assessment]: This session will include a review of therapeutic gains/relapse prevention/assessments.

Visit 16: Post-Treatment Behavioral Tests and MR Scan: This visit will be very similar to Visit 2. Participants will participate in the same type of task inside the MR scanner, while the study staff measures reaction time and psychophysiological responding and brain activation. Participants will view the same images he or she did previously, and may experience the same aversive stimulus as during Visit 2. Participants will again be asked to rate how much they expect to experience the aversive stimulus after each image and will also be asked to report their level of anxiety on a scale from 0 to 100.

Visit 17: Post-Treatment Behavioral Tests and MR Scan: This visit will be very similar to Visit 3. Participants will participate in the same type of task inside the MR scanner, while the study staff measures reaction time and psychophysiological responding and brain activation. Participants will view the same images he or she did previously, and may experience the same aversive stimulus as during Visit 3. Participants will again be asked to rate how much they expect to experience the aversive stimulus after each image and will also be asked to report their level of anxiety on a scale from 0 to 100.

Visit 18: 3-Month Follow-Up Treatment Assessment: This session is similar to Visit 15 and will include review of therapeutic gains/relapse prevention/assessments.

ELIGIBILITY:
Inclusion Criteria:

* Between ages 18-60
* Willing and able to consent to study
* Generally medically and neurologically healthy (including no evidence of intellectual disability or serious cognitive impairment that would interfere with task performance)
* Exposure to Criterion A stressor defined by CAPS-5 and identified by Life Events Checklist-5 (LEC-5)
* Significant PTSD severity as indicated by CAPS-5 diagnosis and/or score >= 25 of at least one month prior to study entry, PTSD is patient's primary concern

Exclusion Criteria:

* Positive urine pregnancy test prior to fMRI, self-reported current pregnancy during screening, or planning pregnancy
* Currently breastfeeding/ lactating
* MRI contraindications (e.g., ferrous metal in head/body)
* Pervasive development disorder history
* Traumatic brain injury (TBI) with current cognitive impairment related to TBI
* Risk of harm to self or others that requires immediate intervention
* Presence of contraindications, current or past allergic or adverse reaction, or known sensitivity to cannabinoid-like substances (dronabinol/marijuana/cannabis/THC, cannabinoid oil, sesame oil, gelatin, glycerin, and titanium dioxide)
* Lack of fluency in English
* Inability to tolerate small, enclosed spaces without anxiety (e.g. claustrophobia
* Exclusively left-handed (score of -100 on Handedness Questionnaire)
* Current or past diagnosis of bipolar, schizophrenia spectrum, psychotic and related disorders
* Current severe alcohol or substance use
* Comorbid mood or anxiety disorder that is primary to PTSD
* Concomitant treatment with medication taken daily that has level 1 evidence indicating severe drug-drug interactions with dronabinol

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Brain Measures | Through study completion, an average of 3 months.
  functional magnetic resonance imaging (fMRI) blood oxygen level-dependent (BOLD) percent signal change within region of interests [amygdala; ventromedial prefrontal cortex; hippocampus]
Psychophysiology | Through study completion, an average of 3 months.
  Skin conductance response (SCR): change in SCR [peak amplitude from 0.5-4.5 sec following stimulus presentation minus average 2 second baseline prior to stimulus presentation].
Expectancy Ratings | Through study completion, an average of 3 months.
  To assess the change in expected likelihood that an aversive cue (e.g. noise burst or shock) will occur or not based on while slide was shown, participants will repeatedly rate their expectancy of the aversive cue using a button box on a scale from 1 to 3 [1 = certain that the aversive cue will be presented; 2 = certain that the aversive cue will not be presented; 3 = uncertain whether the aversive cue will be presented].
PTSD Checklist (PCL-5) | Through study completion, an average of 3 months.
  To track PTSD symptom change for each participant. The PCL-5 is a 20-item questionnaire. The self-report rating scale is 0-4 for each symptom: "Not at all," "A little bit," Moderately," "Quite a bit," and "Extremely", respectively. A total symptom severity score (range - 0-80) can be obtained by summing the scores for each of the 20 items.
Clinician Administered PTSD Scale for Diagnostic and Statistical Manual (DSM)-5 (CAPS-5) | Through study completion, an average of 3 months.
  To track PTSD symptom change for each participant. The CAPS is the gold standard in PTSD assessment. The CAPS is a 30-item structured interview. In addition to assessing the 20 DSM-5 PTSD symptoms, questions target the onset and duration of symptoms, subjective distress, impact of symptoms on social and occupational functioning, improvement in symptoms since a previous CAPS administration, overall response validity, overall PTSD severity, and specifications for the dissociative subtype. The assessor combines information about frequency and intensity of an item into a single severity rating. Total symptom severity score is calculated by summing severity scores for the 20 DSM-5 PTSD symptoms. The five-point CAPS-5 symptom severity rating scale is used for all symptoms (0, Absent; 1, mild; 2, Moderate/threshold; 3, Severe/markedly elevated; 4, Extreme/incapacitating). Total CAPS-5 symptom severity scores range from 0-80, with higher scores indicating worse PTSD symptom severity.
Subjective Units of Distress Scale (SUDS) | Through study completion, an average of 3 months.
  To assess the change in level of distress from 0 to 100 when facing fears. The higher the number on the scale the more severe the level of distress experienced.

SECONDARY OUTCOMES:
Visual Analogue Scale of Mood (VAS) | Through study completion, an average of 3 months.
  Subjective ratings of mood and drug effects on a 0-100. Higher numbers on the scale reflect stronger experiences of different mood and drug effects. Each item is scored individually. There is no overall score.
Drug Effects Questionnaire (DEQ) | Through study completion, an average of 3 months.
  Subjective ratings of drug effects on from 1-5 on the following scales: "Feel", "High", and "Like".
Addiction Research Center Inventory (ARCI) | Through study completion, an average of 3 months.
  A standardized questionnaire of 53 statements for assessing subjective effects of psychoactive drugs. Used to differentiate drug effects from placebo. Participants rate "true" if the statement applies to them or "false" if it does not apply. Specific statements are related to a particular drug class and for that drug class all "true" responses are summed for a total score in that drug class. Higher scores means higher subjective drug effects for particular drug classes. The scales are the Morphine-Benzedrine (score range: 0-16; drug-induced euphoria), Amphetamine (score range: 0-11; specific for dose-related effects of d-amphetamine), Benzedrine (score range: 0-13; an amphetamine scale relating to intellectual efficiency and energy); Pentobarbital-Chlorpromazine (score range: 0-15; sedation); Lysergic Acid (score range: 0-13; dysphoria and somatic symptoms); and Marijuana (score range: 0-12; marijuana's effects).
State-Trait Anxiety Inventory (STAI) | Through study completion, an average of 3 months.
  Measures of state and trait anxiety. The STAI has 20 items for assessing trait anxiety and 20 for state anxiety. State anxiety items include: "I am tense; I am worried" and "I feel calm; I feel secure." Trait anxiety items include: "I worry too much over something that really doesn't matter" and "I am content; I am a steady person." All items are rated on a 4-point scale (e.g., from "Almost Never" to "Almost Always"). The numerical ratings for each of the 20 items assessing trait anxiety are summed for a total trait anxiety score. The numerical ratings for each of the 20 items assessing state anxiety are summed for a total state anxiety score. Scores on the trait and state anxiety scales of the STAI can range from 20-80. STAI scores are commonly classified as "no or low anxiety" (scores 20-37), "moderate anxiety" (scores 38-44), and "high anxiety" (scores 45-80).
End of Session Questionnaire (ESQ) | Through study completion, an average of 3 months.
  Includes 5 questions total. The first two question ask the participant to select one of several statements that best describes the effect of the capsule they took during that visit. The second question asks the participant to guess what they thought they received in the capsule and how confident they are. The third question asks the participant to rate how much the liked or disliked the effects of the capsule overall on a scale from -5 to 5, with -5 being "disliked a lot", 0 being "neutral", and 5 being "liked a lot". The fourth question asks participants to check "yes" or "no" if they would take the capsule again. Finally, the last question is a free text response asking the participant if they experienced any unusual reactions or if they have any comments or observations that may be relevant to the study.
Heart Rate | Through study completion, an average of 3 months.
  Heart rate
Blood Pressure | Through study completion, an average of 3 months.
  Systolic and diastolic blood pressure will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Christine A Rabinak, PhD, Principal Investigator — Wayne State University
Locations (1):
- Eugene Applebaum College of Pharmacy and Health Sciences, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rabinak CA, Kilgore PE, Lumley MA, Rauch SAM. Randomized trial of delta-9-tetrahydrocannabinol (THC) versus placebo to augment the effects of prolonged exposure therapy on fear extinction learning in post-traumatic stress disorder: Study rationale and protocol. Contemp Clin Trials. 2026 Jan;160:108148. doi: 10.1016/j.cct.2025.108148. Epub 2025 Nov 19. PMID 41270825